CLINICAL TRIAL: NCT01041001
Title: Randomized, Open-Label, Multi-Center and Phase 3 Clinical Trial to Compare the Efficacy and Safety of Cartistem® and Microfracture in Patients With Knee Articular Cartilage Injury or Defect
Brief Title: Study to Compare Efficacy and Safety of Cartistem and Microfracture in Patients With Knee Articular Cartilage Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-CRP-005
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2012-04

CONDITIONS: Cartilage Injury; Osteoarthritis
Keywords: Umbilical Cord Blood; Mesenchymal Stem Cells; cartilage injury; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cartistem (Experimental): A single dose of 500㎕/㎠ of cartilage defect
  Interventions: Biological: Cartistem
- Microfracture treatment (Active Comparator)
  Interventions: Procedure: Microfracture treatment

INTERVENTIONS:
Biological: Cartistem — allogeneic-unrelated umbilical cord blood-derived mesenchymal stem cell product
  Arms: Cartistem
Procedure: Microfracture treatment
  Arms: Microfracture treatment

SUMMARY:
The purpose of the study is to assess and compare the safety and efficacy of the allogeneic-unrelated umbilical cord blood-derived mesenchymal stem cell product (Cartistem®) to that of a microfracture treatment in patients with articular cartilage defect or injury.

DETAILED DESCRIPTION:
The cartilage is a unique avascular, aneural tissue that does not regenerate easily once damaged. Chondral defects or damages to articular cartilages due to accidents, necrosis of subchondral bone tissue, or arthritis have become some of the more common disorders today. About 15% of the world's population is reportedly suffering from cartilage and joint damages such as degenerative arthritis and rheumatoid arthritis. As population aging progresses and as more young people start taking up active sports, the size of the target patient group is also growing. However, despite ongoing research, an effective treatment for cartilage defects is yet to be discovered. Various different types of treatments are currently in use, such as drug therapy, arthroscopy, and artificial joint surgery. However, they all fail to address the root cause. Complete treatment, or regeneration of damaged or defective cartilage is impossible and continuous drug administration or secondary surgeries are required in many cases.

As a way of regenerating the damaged or defective cartilage tissue, treatment of localized damage to articular cartilage using autologous chondrocytes is currently under review. A few life science companies both home and abroad are marketing this method of treatment called 'autologous chondrocyte transplant'. The treatment involves the extraction of healthy cartilage tissue from the patient which is then cultured and transplanted into the damaged site.

However, this treatment requires the extraction of chondrocytes directly from the patient and thus causes trauma in healthy articular cartilage. Also, this type of treatment cannot be applied to large lesions, nor is the efficacy satisfactory in patients over the age of 40 whose cellular activation levels are low. Thus, autologous chondrocyte transplant is rather limited in the number of cells harvested and their activation level and is therefore restricted in terms of treatment site, severity of the condition, and the size of lesion. The current technology allows the application of treatments in local cartilage defects but not in degenerative arthritis or rheumatoid arthritis. The technology needs to be taken up to another level in order to benefit such prevalent arthritic disorders. Treatments using stem cells do not cause damage to healthy articular cartilage as they don't require the harvesting of healthy cartilage tissues from the patients. Moreover, the number of successfully cultured cells is larger due to the excellent proliferation capability of stem cells and thus, mass supply is possible.

This clinical trial for the stem cell therapies is essential because treatment of cartilage defects with umbilical cord blood-derived mesenchymal stem cells, known to have the highest level of activity among all adult stem cells, opens the possibility of articular cartilage regeneration even for aged patients and patients with large lesions unable to benefit from existing treatments.

The biggest challenge faced by nations competing in the field of "tissue differentiation and regeneration using stem cells" is the question of whether or not the use of embryonic stem cells is ethical. Chondrogenesis using umbilical cord blood-derived mesenchymal stem cells can not only avoid similar challenges, but also present an innovative treatment mode with significant clinical implications for the patients.

In the clinical study, mesenchymal stem cells will be isolated from umbilical cord blood and cultured, mixed with semi- solid polymer, and administered into the cartilage tissue lesion by orthopedic surgery in order to stimulate the regeneration of defective cartilage tissue and to improve their functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee joint cartilage defect or injury of ICRS (International Cartilage Repair Society) Grade 4 confirmed by arthroscopy (At screening, patients diagnosed as such with an MRI may be included)
* Male or female patients at least 18 years of age
* Patients whose lesion (unilateral joint) is 2 ㎠ ~ 9㎠ in size
* Patients with articular swelling, tenderness and active range of motion of Grade 2 or below
* Patients with pain in affected joint of 60-mm or below on a 100-mm VAS (visual analogue scale)
* Patients with adequate blood coagulation activity, PT(INR) < 1.5, APTT <1.5×control
* Patients with adequate renal function, Creatinine ≤ 2.0 ㎎/㎗, levels of proteinuria measured with Dipstick: trace or less
* Patients with adequate hepatic function, Bilirubin ≤ 2.0 ㎎/㎗, AST/ALT ≤ 100 IU/L
* Patients who have received no surgery or radiation therapy in the affected joint within the past 6 six weeks, and have recovered from the side effects of such past treatments
* Female patients of childbearing potential must agree to practice adequate methods of birth control to prevent pregnancy during the study
* Patients whose physical examination results show no ligament instability of Grade II or above (Grade 0: none, Grade I: 0-5 mm, Grade II: 5-10 mm, Grade III: >10 mm)
* Patients who voluntarily agreed to enroll in the study and signed an informed consent form

Exclusion Criteria:

* Patients with autoimmune disease or the medical history
* Patients with infections requiring parenteral administration of antibiotics
* Patients with myocardial infarction, ischemic heart failure, other serious heart conditions or uncontrolled hypertension, or any medical history of such diseases
* Patients with serious internal diseases
* Patients who are currently pregnant or nursing
* Patients with psychotic diseases, epilepsy, or any history of such diseases
* Patients with alcohol abuse
* Patients who smoke excessively
* Patients with chronic inflammatory articular diseases such as rheumatoid arthritis
* Patients who were enrolled in any other clinical trials within the past four weeks
* Patients who had been administered with immunosuppressants such as Cyclosporin A or azathioprine within the past six weeks
* Patients whose physical examination results show ligament instability of Grade II or above (Grade 0: none, Grade I: 0-5 mm, Grade II: 5-10 mm, Grade III: >10 mm)
* Patients with a known history of hypersensitivity/allergy to gentamicin
* Patients who the principal investigator considers inappropriate for the clinical trial due to any other reasons than those listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
ICRS Cartilage Repair Assessment will follow to determine the appropriate grade. The treatment will be considered efficacious if the ICRS grade drops by at least 1 grade or more from baseline to week 48. | Week 0 and 48

SECONDARY OUTCOMES:
Degree of improvement in the grade of joint pain measured on a 100-mm VAS (Visual Analogue Scale) | Week 0, 2, 4, 8, 12, 24, 36 and 48
Grade of cartilage regeneration in patients who agreed to a biopsy during arthroscopy at week 48 | Week 48
Changes in WOMAC scores | Week 0, 2,4,8,12,24,36 and 48
Changes in IKDC Subjective Score | Week 0, 2, 4, 8, 12, 24, 36 and 48
ICRS scores | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Hong-chul Lim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (8):
- South Korea (8):
  - Gachon University Gil Hospital, Incheon, Gyunggido
  - Inha University Hospital, Incheon
  - Hanyang University Medical Center, Seoul
  - Seoul Veterans Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim HC, Park YB, Ha CW, Cole BJ, Lee BK, Jeong HJ, Kim MK, Bin SI, Choi CH, Choi CH, Yoo JD; Cartistem Research Group; Yoon JR, Chung JY. Allogeneic Umbilical Cord Blood-Derived Mesenchymal Stem Cell Implantation Versus Microfracture for Large, Full-Thickness Cartilage Defects in Older Patients: A Multicenter Randomized Clinical Trial and Extended 5-Year Clinical Follow-up. Orthop J Sports Med. 2021 Jan 12;9(1):2325967120973052. doi: 10.1177/2325967120973052. eCollection 2021 Jan. PMID 33490296